CLINICAL TRIAL: NCT02998606
Title: Movantik for Opioid-Related Esophageal Disorders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator left Institution
Sponsor: Temple University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23289
Record Dates: First submitted 2016-12-14; First posted 2016-12-20 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Opioid-Induced Disorders; Esophagus Disorder
MeSH Terms: conditions — Esophageal Diseases | interventions — naloxegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group (Experimental): MOVANTIK™ (Naloxegol) 25 mg oral capsule, daily
  Interventions: Drug: Naloxegol
- Control Group (Placebo Comparator): Placebo Oral Capsule 25 mg, daily
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Naloxegol — MOVANTIK™ 25 mg, daily
  Other Names: Movantik
  Arms: Study Group
Drug: Placebo Oral Capsule — Placebo 25 mg, daily
  Other Names: Placebo
  Arms: Control Group

SUMMARY:
To date, few studies have assessed the effect of opioids on esophageal motility, mostly assessed the effect of single-dose intravenous morphine on esophageal motility. Recently a large retrospective study assessing the effect of opioids on esophageal motility found that esophageal motor dysfunction are common in chronic opioid users whether studied on opioids and off opioids. In addition, current opioid users also had significantly higher integrated relaxation pressure and manometric patterns consistent with type III achalasia. (Ratuapli 2015) Peripherally acting mu opioid receptor antagonists (PAMORA) appear to be useful to reduce the peripheral effects of mu opioid receptor agonists to delay gastrointestinal transit without affecting the centrally mediated analgesic effects. MOVANTIK™ (Naloxegol) is the first oral peripherally acting mu opioid receptor antagonists for opioid-induced constipation. MOVANTIK™ (Naloxegol) has been recently approved for opioid-induced constipation. Given orally, 25 mg daily it improves symptoms of constipation. At this dose, MOVANTIK™ (Naloxegol) is effective and safe, with a limited side effect profile and is associated with preservation of centrally mediated analgesia.

This study will explore the safety and tolerability of MOVANTIK™ (Naloxegol) in this patient population.

The investigational hypothesis is that MOVANTIK™ (Naloxegol) could improve opioid- induced esophageal motility disorders

DETAILED DESCRIPTION:
Background MOVANTIK™ (Naloxegol) can alleviate the adverse effects associated with frequent opiate use. The GI system is a common site for their unintended effects of opiate use, but literature suggests that peripherally acting opioid agonist may provide relief in the instance of GI dysfunction. (Holzer 2007) Toxicology and pharmacology summary

14 Phase I studies were completed with 439 health volunteers participating. MOVANTIK™ (Naloxegol) has been tested in a standard range of safety pharmacology studies including an absorption, distribution, metabolism and excretion study, a QTc (corrected QT interval) study, several PK (pharmacokinetic) studies, and a study to determine its central and peripheral pharmacodynamics effects. MOVANTIK™ (Naloxegol) is metabolized primarily by cytochrome P450 enzyme (CYP)-3A4 and CYP3A5 and is a substrate for a P-glycoprotein transporter. Drug-drug interaction studies were performed for a strong and a moderate CYP3A4 inhibitor, a CYP3A5 inhibitor and P-glycoprotein transporter inhibitor.

Clinical Safety summary MOVANTIK™ (Naloxegol) was initially tested in 439 healthy volunteers across 14 Phase I studies. Ascending-dosing studies were performed with first dose ranging from 8-1000 mg, followed by twice daily dosing ranging from 25-250 mg, all administered intravenously. Another ascending dose study was completed in older volunteers (age 65 and older) in Japan to determine the effects of advanced age on PK values. Phase IIb and II studies exposed 1497 patients to dosages ranging from 5 mg to 50 mg for periods of time varying from 24 to 52 weeks. MOVANTIK™ (Naloxegol) has shown acceptable safety profile and was well-tolerated at 5 mg and 25 mg. The 50 mg cohort had shown increased frequency of GI adverse events (abdominal pain, nausea and diarrhea) when compared to the 25 mg and 5 mg cohorts. The 25 mg dose was the maximum used across the 5 phase III studies. Two 12 week placebo-controlled double-blind studies were completed to confirm safety and efficacy, as well as a 12 week double-blind safety extension, a randomized 52-week open-label parallel group, long-term safety study and a placebo-controlled, double-blind study in patients with cancer-related pain. The efficacy studies demonstrated the therapeutic effect of MOVANTIK™ (Naloxegol) was independent of age, gender, race, body mass index, region, use of anticholinergics, response to previous laxative use, type of opioid, or dose of opioid. Phase III studies demonstrated that MOVANTIK™ (Naloxegol) is generally safe and well tolerated at doses up to 25 mg once daily in patients with OIC (opioid-induced constipation) up to 52 weeks of treatment.

Acute and chronic use of opioids is associated with a variety of adverse effects on the gastrointestinal tract. The effect of opioids on gastric, small bowel, and colonic motility has been well characterized. The main esophageal abnormalities seen were impaired LES (lower esophageal sphincter) relaxation. Recently a large retrospective study assessing the effect of opioids on esophageal motility using, for the first time, HREM and the Chicago classification of esophageal motility disorders v3.0 found that Esophageal motor dysfunction are common in chronic opioid users whether studied on opioids and off opioids. (K raichely 2010) However, opioid use within 24 h of manometry was associated with increased EGJ ( Esophagogastric junction) outflow obstruction and other spastic esophageal motor abnormalities. In addition, current opioid users also had significantly higher integrated relaxation pressure and manometric patterns consistent with type III achalasia.

Benefit/risk and ethical assessment Preliminary data suggests a relationship between opioid use and esophageal dysfunction. The decline in quality of life associated with esophageal disorders may discourage patients from taking opioids, subjecting them to unwarranted pain. MOVANTIK™ (Naloxegol) is an opioid antagonist specifically designed to work outside of the central nervous system. This allows relief from undesired peripheral effects of opioids without disrupting analgesic effects. The use of MOVANTIK™ (Naloxegol) has the potential to mediate esophageal dysfunction while preserving vital pain relief.

Patients for whom MOVANTIK™ (Naloxegol) is contraindicated will be excluded as well as those taking strong CYP3A4 inhibitors or strong CYP3A4 inducers and other opioid antagonists. In the Phase III studies, adverse events of abdominal pain (21% v 7%), diarrhea (9% v 5%), nausea (8% v 5%), flatulence (6% v 3%), vomiting (5% v 4%), headache (4% v 3%), and hyperhidrosis (3% v <1%) were observed at greater rates among the 25 mg cohort when compared to placebo.. The current study is designed to explore the potential benefit or effect of Naloxegol on upper GI motility and clinical symptoms inpatients receiving opioid

Study design This is a single center, randomized, placebo-controlled, double-blind study to determine the effect of MOVANTIK™ (Naloxegol) on opioid-related esophageal motility disorders.

This study consists of 2 week screening period, a 4 week treatment period and a 2 week follow-up period. Eligible patients will be placed in either a study group or a control group, with 15 patients in each study arm. Patients will receive a High Resonance Esophageal Manometry (HREM) at Visits 2 and 3.

Visit one (Day -14) Patients will be seen and informed consent will be obtained. Inclusion and exclusion criteria will be review to determine eligibility.

At visit 1 the following procedures will be performed:

* Obtain demographic, endoscopic, clinical, and prior manometric data to determine eligibility
* Review medication history
* Physical Examination
* Obtain Weight and Height
* Obtain Seated Vital Signs (Includes Oral temperature, Pulse, BP and respiratory rate)
* Collect blood sample for Serum Pregnancy Test1
* Patients complete the following questionnaires

  o Patient Assessment of GI Symptoms (PAGI-SYM)
* Patients will be given a daily diary to complete throughout the next two weeks.

Visit two (Day 0 ± 3 days) Patients will return to clinic after fasting2, except for medications with water in the morning, and will undergo a HREM. Review the daily diary, manometric and the inclusion/exclusion criteria to determine eligibility. The following procedures will occur before the patient receives study drug. After the procedure, patients will be started on the study drug (Movantik 25 mg) or Placebo daily on a random double blind basis.

At visit 2 the following procedures will be performed:

* Review and record adverse event which have occurred from the signing of the ICF (informed consent form) to Visit 2
* Review concomitant medications and Daily diary
* Obtain Weight and Height
* Obtain Seated Vital Signs (Includes Oral temperature, Pulse, BP and respiratory rate)
* Patients complete the following questionnaires

  * Patient Assessment of GI Symptoms (PAGI-SYM)
  * Lower GI symptoms questionnaire
  * McGill Pain inventory
  * SF-36
  * Chest pain symptom questionnaire
  * GERD (gastroesophageal reflux disease) symptom check list
* Patients will undergo a HREM
* Obtain study number, randomize patients and dispense investigational product.

Visit Three (Day 2± 3 days) Patients will receive a phone call to assess their initial response to treatment two days after they start the study drug and better assess the safety of the drug.

During Visit 3the following procedures will be performed:

* Review and record adverse event which have occurred from the signing of the ICF to Visit 3
* Review concomitant medications

Visit four (Day 28 ± 3 days)

* Review and record adverse event which have occurred from Visit 3 to Visit 4
* Review concomitant medications and Daily diary
* Obtain Weight and Height
* Obtain Seated Vital Signs (Includes Oral temperature, Pulse, BP and respiratory rate)
* Patients complete the following questionnaires

  * Patient Assessment of GI Symptoms (PAGI-SYM)
  * Lower GI symptoms questionnaire
  * McGill Pain inventory
  * SF-36
  * Chest pain symptom questionnaire
  * GERD symptom check list
* Patients will undergo a HREM2 (High Resonance Esophageal Manometry)
* Perform investigational product accountability.

Visit five (Day 42 ± 7 days) Patients will be seen to ensure collection of the daily diaries and for a final safety assessment

* Review and record adverse event which have occurred from Visit 4 to Visit 5 and further detail any adverse event that have occurred throughout the study
* Review concomitant medications and return daily diary
* Obtain Weight and Height
* Obtain Seated Vital Signs (Includes Oral temperature, Pulse, BP and respiratory rate)

Early Withdrawal/Early Termination

Patients who withdraw early will be encouraged to complete their Visit 3 requirements:

* Review and record adverse event which have occurred from Visit 2 to withdrawal (termination) date
* Review concomitant medications and Daily diary
* Obtain Weight and Height
* Obtain Seated Vital Signs (Includes Oral temperature, Pulse, BP and respiratory rate)
* Patients complete the following questionnaires

  * Patient Assessment of GI Symptoms (PAGI-SYM)
  * Lower GI symptoms questionnaire
  * McGill Pain inventory
  * SF-36
  * Chest pain symptom questionnaire
  * GERD symptom check list
* Perform investigational product accountability

Rationale for study design, doses and control groups This study seeks to determine the effectiveness of MOVANTIK™ (Naloxegol) in treating patients with opioid-induced esophageal disorders. MOVANTIK™ (Naloxegol) has already been shown to be effective in other opioid induced gastric disorders. To the Investigator's knowledge there has been no double-blind randomized control trial evaluating the effects of MOVANTIK™ (Naloxegol) on opioid induced-esophageal disorders. The same dosage that has been proven effective in other patient populations will be used. The use of a control group eliminates potential bias in the patient-reported outcome endpoints. The enrollment goal is 50 patients for this study. A recent study showed all 15 enrolled patients showed signs of opioid-induced motility abnormalities on HREM. (Kraichely 2010) Relatively large effects can be expected in this sample size. Using G* power 3 will ensure that that a sample size of 42 patients will give provide a 95% chance of detecting a large effect size (defined as 0.80 population s.d. between groups) between the two groups as significant at the 5% level (two tailed) using t -test between means. Enrolling 50 patients ensures an adequate amount of patients complete the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Age 18-85, Males and Females
3. On a stable daily opioid dose for various indications for at least 4 weeks prior to the HREM (High Resonance Esophageal Manometry
4. Symptoms of odynophagia, dysphagia, or chest pain based on symptoms recorded on the PAGI-SYM

Exclusion Criteria:

1. Renal impairment (cct<60) or severe Hepatic impairment as defined by the Child-Pugh Classification (Appendix J)
2. Concomitant use of strong or moderate CYP3A4 inhibitors, strong CYP3A4 inducers, NSAIDS, Plavix/Clopidogrel and other opioid antagonists
3. History of GI obstruction, bowel perforation, or with potential for either based on investigator's clinical judgment
4. Subjects with known Barrett's esophagus or peptic stricture on endoscopy
5. Subjects with previous upper gastrointestinal surgery
6. Pregnant, plan to be pregnant, or are breastfeeding
7. Women of childbearing potential who are unwilling to use contraceptives throughout the course of treatment
8. Subjects with serious co-morbidities (Cardiovascular, respiratory, renal, hepatic, hematologic, endocrine, neurologic) which may prevent the patient to participate in the study based on PI's clinical judgment or malignancy
9. Patients with an increased risk of gastrointestinal perforation due to conditions that may be associated with localized or diffuse reduction of structural integrity in the wall of the gastrointestinal tract (e.g. peptic ulcer disease, Ogilvie's syndrome, diverticular disease, infiltrative gastrointestinal tract malignancies or peritoneal metastases).
10. Subjects with upper airway symptoms (such as hoarseness, wheezing or laryngospasm)
11. Patients taking baclofen or sucralfate and those unwilling to discontinue prohibited medications.
12. Known history of substance abuse
13. Subject unable to consent or is unwilling to provide informed consent
14. History of major comorbid psychiatric conditions including mania and schizophrenia or severe current depression
15. At-risk populations, including prisoners and mentally challenged. Any condition or is in a situation which may put him/her at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study (e.g., difficulty hearing, cognitive impairment)
16. Known allergy to MOVANTIK™ (Naloxegol)
17. Patients with a history of cancer within past 5 years prior to the screening visit
18. Patients with a medical condition which may disrupt the blood-brain barrier

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-01; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Manometric improvement in IRP (Integrated Relaxation Pressure) | 28 days
  The effect of MOVANTIK™ (Naloxegol) on motor function, categorized as a 25% (mmHg) improvement in IRP (Integrated Relaxation Pressure) on high resolution esophageal manometry from baseline to visit three, comparing study group to placebo control group.

SECONDARY OUTCOMES:
Overall Symptom Management | 28 days
  Mean change from baseline to visit three in subject esophageal symptom scores according to the PAGI-SYM.
Pain Management | 28 days
  Mean change from baseline to visit three in subject esophageal symptom scores according to the McGill pain inventory.
GERD Symptom Management | 28 days
  Mean change from baseline to visit three in subject esophageal symptom scores according to the GERD symptom check list.
Chest Pain Management | 28 days
  Mean change from baseline to visit three in subject esophageal symptom scores according to the chest pain symptom questionnaire.
Daily Symptom Management | 28 days
  Mean change from baseline to visit three in subject esophageal symptom scores according to the daily diary
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability | 42 days
  The occurrence of adverse events and early withdrawal in study group when compared to placebo control group to determine safety and tolerability.
Quality of Life | 28 days
  Mean change in patient-reported quality of life according to the SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Ron Schey, MD, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holzer P. Treatment of opioid-induced gut dysfunction. Expert Opin Investig Drugs. 2007 Feb;16(2):181-94. doi: 10.1517/13543784.16.2.181. PMID 17243938
- [Background] Ratuapli SK, Crowell MD, DiBaise JK, Vela MF, Ramirez FC, Burdick GE, Lacy BE, Murray JA. Opioid-Induced Esophageal Dysfunction (OIED) in Patients on Chronic Opioids. Am J Gastroenterol. 2015 Jul;110(7):979-84. doi: 10.1038/ajg.2015.154. Epub 2015 Jun 2. PMID 26032150
- [Background] Mittal RK, Frank EB, Lange RC, McCallum RW. Effects of morphine and naloxone on esophageal motility and gastric emptying in man. Dig Dis Sci. 1986 Sep;31(9):936-42. doi: 10.1007/BF01303214. PMID 3731985
- [Background] Penagini R, Bartesaghi B, Zannini P, Negri G, Bianchi PA. Lower oesophageal sphincter hypersensitivity to opioid receptor stimulation in patients with idiopathic achalasia. Gut. 1993 Jan;34(1):16-20. doi: 10.1136/gut.34.1.16. PMID 8381758
- [Background] Penagini R, Picone A, Bianchi PA. Effect of morphine and naloxone on motor response of the human esophagus to swallowing and distension. Am J Physiol. 1996 Oct;271(4 Pt 1):G675-80. doi: 10.1152/ajpgi.1996.271.4.G675. PMID 8897888
- [Background] Dowlatshahi K, Evander A, Walther B, Skinner DB. Influence of morphine on the distal oesophagus and the lower oesophageal sphincter--a manometric study. Gut. 1985 Aug;26(8):802-6. doi: 10.1136/gut.26.8.802. PMID 4018646
- [Background] Penagini R, Bianchi PA. Effect of morphine on gastroesophageal reflux and transient lower esophageal sphincter relaxation. Gastroenterology. 1997 Aug;113(2):409-14. doi: 10.1053/gast.1997.v113.pm9247457.
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Kraichely RE, Arora AS, Murray JA. Opiate-induced oesophageal dysmotility. Aliment Pharmacol Ther. 2010 Mar;31(5):601-6. doi: 10.1111/j.1365-2036.2009.04212.x. Epub 2009 Dec 8. PMID 20003176
- [Background] Conklin JL. Evaluation of Esophageal Motor Function With High-resolution Manometry. J Neurogastroenterol Motil. 2013 Jul;19(3):281-94. doi: 10.5056/jnm.2013.19.3.281. Epub 2013 Jul 8. PMID 23875094